CLINICAL TRIAL: NCT04709016
Title: The Use of Chemsex (Drug Use in a Sexual Context) Among MSM (Men Who Have Sex With Men) and Transgender People in France, Whether or Not Taking PrEP, and Its Impact on PrEP Adherence
Brief Title: Drug Use During Sex and Its Impact on Taking PrEP (Pre-Exposure Prophylaxis) : CONSUME
Acronym: CONSUME
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02182-37
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-05

CONDITIONS: Drug Dependence
Keywords: Chemsex; PrEP
MeSH Terms: conditions — Substance-Related Disorders; Chemsex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- male or transgender patients: of sexual orientation MSM (men having sex with men) or bi-sexual, consultant in sexual health centers
  Interventions: Behavioral: self-questionnaire

INTERVENTIONS:
Behavioral: self-questionnaire — self-questionnaire assessing Chemsex's (drug use in a sexual context) consumption over the last 12 months

SUMMARY:
This is a cross-sectional, single-center observational study conducted from October 2020 to March 2021 in Ile de France at the infectious disease of CHU Bichat (PrEP and CeGIDD(Free Center for Information, Screening and Diagnosis of Infections by Human Immunodeficiency Viruses, Viral Hepatitis and Sexually Transmitted Infections) consultation). It concerns adult subjects of male or transgender sex, of MSM (men having sex with men) or bi-sexual orientation. The data are collected by self-questionnaire evaluating the consumption of Chemsex (drug use in a sexual context) over the last 12 months, the existence or not of addiction treatment, the history of STIs (sexually transmitted infections) and adherence to PrEP (for subjects taking PrEP) during the last sexual intercourse (ANRS questionnaire, used in the PREVENIR study).

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* male or transgender
* MSM or bi-sexual orientation
* adult consultant at Bichat Hospital (CeGIDD or PrEP consultation)
* adult with a Smartphone (online self-questionnaire)

Exclusion Criteria:

* For the group "taking PrEP": adult taking PrEP for less than 3 months
* Refusal of participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male or transgender MSM or bi-sexual orientation
Study Population: The study concerns subjects of male or transgender sex, of MSM or bi-sexual sexual orientation, consulting in sexual health centers.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
compare in an MSM and transgender population, the use of Chemsex depending on whether or not PrEP is taken | inclusion

SECONDARY OUTCOMES:
Reported adherence to PrEP | inclusion
The existence or not of psychological comorbidity and the existence of addictological care | inclusion
The number of sexually transmitted infections at inclusion | inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- SMIT - Hôpital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: No